CLINICAL TRIAL: NCT05473637
Title: Deciphering, Construction and Validation of Magnetic Resonance Imaging Maps, Clinical Features and Outcomes in Genetic and Nongenetic Cerebral Small Vessel Diseases
Brief Title: Taiwan Associated Genetic and Nongenetic Small Vessel Disease
Acronym: TAG-SVD
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201911029RINB
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Small Vessel Diseases; Cadasil; HTRA1-Related Autosomal Dominant Cerebral Angiopathy; COL4A1-Related Brain Small Vessel Disease With Haemorrhage; Fabry Disease; Magnetic Resonance Imaging; Next-generation Sequencing; Stroke
MeSH Terms: conditions — Cerebral Small Vessel Diseases; CADASIL; Fabry Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Each patient had a blood sample collected, and their DNA was extracted and sent for next-generation sequencing (NGS) with probes designed to target five candidate CSVD genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genetic group: Patients who have positive DNA results by NGS screening of the following 5 genes: NOTCH3 (19q13.12), HTRA1 (10q26.13), GLA (Xq22.1), TREX1 (3p1.31) and COL4A1 (13q34).
  Interventions: Diagnostic Test: MRI
- Nongenetic group: Patients who have negative DNA results by NGS screening .
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Patients will repeat study-protocol MRI at baseline (enrollment) and at least once in 1 year or 2 years follow-up (depends on availability).

SUMMARY:
The TAG-SVD enrolled patients with clinical and neuroimaging features of cerebral small vessel disease (CSVD). All enrolled patients will receive next-generation sequence (NGS) with probes designed to target five candidate CSVD genes, and patients will be divided into genetic or non-genetic groups accordingly. Their clinical features and outcome will be followed for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

Participants must have at least one of the following symptoms/signs or history

* stroke (especially small vessel occlusion type of ischaemic stroke, spontaneous ICH or young stroke)
* cognitive impairment or dementia
* gait disturbance
* parkinsonism (especially vascular parkinsonism features)
* headache (especially migraine)
* positive family history of hereditary CSVD
* MRI evidence of CSVD (MRI may be done for other reasons), including mild to moderate white matter hyper intensity, any lacune, or any cerebral microbleed

Exclusion Criteria:

* MRI evidence of CSVD due to other inflammatory, malignancy, or structural lesions
* patients or family members not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients with clini-cal and neuroimaging features of CSVD in the neurology outpatient clinic of National Taiwan University Hospital. The clinical features for being enrolled in the TAG-SVD cohort included stroke (especially small vessel occlusion type of ischaemic stroke, spontaneous ICH or young stroke), cognitive impairment, gait disturbance, parkinsonism, headache or a positive family history of hereditary CSVD. The neuroimaging features were at least one evident magnetic resonance imaging (MRI) feature of CSVD
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incident stroke | 2 years
  Clinical stroke, including transient ischemic attack, ischemic stroke, or intracerebral hemorrhage.
  The stroke is defined by a focal neurological deficits lasting more than 24 hours, with accompanied neuroimaging evidence of infarct or hemorrhage in corresponding brain area.

SECONDARY OUTCOMES:
Number of patients with incident dementia | 2 years
  Vascular cognitive impairment (VCI), vascular dementia (VaD), or Alzheimer's dementia or Vascular dementia according to latest diagnostic criteria.
  Alzheimer's disease diagnostic criteria: National Institute of Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease (PMID: 21514247)
  Vascular dementia diagnostic criteria: Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data that support the current study are available upon reasonable request to the corresponding author.

REFERENCES:
- [Result] Chen CH, Chu YT, Chen YF, Ko TY, Cheng YW, Lee MJ, Chen PL, Tang SC, Jeng JS. Comparison of clinical and neuroimaging features between NOTCH3 mutations and nongenetic spontaneous intracerebral haemorrhage. Eur J Neurol. 2022 Nov;29(11):3243-3254. doi: 10.1111/ene.15485. Epub 2022 Jul 18. PMID 35781912
- [Result] Zhang R, Chen CH, Tezenas Du Montcel S, Lebenberg J, Cheng YW, Dichgans M, Tang SC, Chabriat H. The CADA-MRIT: An MRI Inventory Tool for Evaluating Cerebral Lesions in CADASIL Across Cohorts. Neurology. 2023 Oct 24;101(17):e1665-e1677. doi: 10.1212/WNL.0000000000207713. Epub 2023 Aug 31. PMID 37652700
- [Result] Shen YC, Chen YF, Cheng YW, Chen CH, Jeng JS, Tang SC. Characteristics and temporal evolution of asymptomatic diffusion-weighted imaging lesions in patients with cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL). Eur J Neurol. 2024 Dec;31(12):e16519. doi: 10.1111/ene.16519. Epub 2024 Oct 11. PMID 39392097
- [Result] Fislage M, Chen CH, Cheng YW, Chen YF, Tang SC. Subcortical volumes and cognition in CADASIL - A pilot study. Cereb Circ Cogn Behav. 2024 Oct 9;7:100371. doi: 10.1016/j.cccb.2024.100371. eCollection 2024. PMID 39493517
- [Result] Cheng YW, Liao YC, Chen CH, Chung CP, Fann CSJ, Chang CC, Lee YC, Tang SC. Contribution of the APOE Genotype to Cognitive Impairment in Individuals With NOTCH3 Cysteine-Altering Variants. J Am Heart Assoc. 2023 Nov 21;12(22):e032689. doi: 10.1161/JAHA.123.032689. Epub 2023 Nov 20. PMID 37982214
- [Result] Lin CW, Yang ZW, Chen CH, Cheng YW, Tang SC, Jeng JS. Reduced macular vessel density and inner retinal thickness correlate with the severity of cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL). PLoS One. 2022 May 26;17(5):e0268572. doi: 10.1371/journal.pone.0268572. eCollection 2022. PMID 35617208